CLINICAL TRIAL: NCT03448237
Title: Remédiation Orthophonique couplée à Une Prise en Charge Proprioceptive de la Dyslexie. Etude Comparative randomisée
Brief Title: Orthophonic and / or Proprioceptive Treatment of Developmental Dyslexia.
Acronym: Pro-Pho-Dys
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Scalab CNRS 9193 (Other)
Responsible Party: Principal Investigator, Luc-Marie Virlet, Coordinating Investigator, Scalab CNRS 9193
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Scalab 2015-024EL; ID RCB : 2015-A01792-47 (Other: ANSM, France)
Record Dates: First submitted 2018-02-15; First posted 2018-02-28 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Developmental Dyslexia
MeSH Terms: conditions — Dyslexia | interventions — Speech Therapy

STUDY DESIGN:
Intervention Model Description: Interventional comparative study over 9 months, of three modes of care: Speech-language, or proprioceptive, or combined (speech therapy or proprioceptive); In view of the lack of recruitment of dyslexic children who had stopped speech therapy, we decided to keep only two comparative arms to our study: of two modes of care: Speech-language, or combined (speech therapy or proprioceptive)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Speech therapy (Active Comparator): Speech therapy adapted to the child,
  Interventions: Other: Speech Therapy
- Combined Treatment (Experimental): Association of speech therapy and proprioceptive treatment, adapted to the child.
  Interventions: Other: Speech Therapy; Other: Proprioceptive treatment

INTERVENTIONS:
Other: Speech Therapy — Speech therapy adapted to the child, at least 25 sessions over 9 months.
  Other Names: Orthophonic treatment
Other: Proprioceptive treatment — Proprioceptive treatment adapted to the child.
  This treatment aims to stabilize a central reference instability revealed to Maddox Postural by the use of neurosensory decoys::
  * Proprioceptive stimulation of oculomotor muscles (active prisms).
  * Oral somatosensory stimulation (ALPH).
  * Proprioceptive antigravity stimulation (proprioceptive sole).
  * Proprioceptive reprogramming exercise.
  Following the teaching of the University Diploma: Perception-Action, Learning Disorders (University of Bourgogne, France)
  Arms: Combined Treatment

SUMMARY:
To show the interest of the association of proprioceptive and orthophonic care of dyslexic children. The assumption is that proprioceptive support by correcting a centrally located spatial localization instability restores the ability to automate.

It allows a gain of effectiveness of the orthophonic remediation of the reading of dyslexic children.

Interventional comparative study over 9 months, of three modes of care: Speech-language, or proprioceptive, or combined (speech therapy or proprioceptive)

ELIGIBILITY:
Inclusion Criteria:

* Developmental dyslexia, (CIM-10)
* Having benefited from 2 years of speech therapy.
* Pathological reading delay of more than 24 months or -2 standard deviations.
* Either in the course of orthophonic care, or having stopped any orthophonic care.

Exclusion Criteria:

* Refractive correction above +/- 1.5 diopters.
* Absence of binocular vision.
* Amblyopia.
* Convulsion.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2018-02-17 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2020-10-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline C index ( Alouatte-R test) at 9 months | Baseline, at nine months
  Number of correctly read words (standard deviation)

SECONDARY OUTCOMES:
Change from baseline TL index ( Alouatte-R test) at 9 months | Baseline, at nine months
  Reading time in second (TL) (standard deviation)
Change from baseline M index ( Alouatte-R test) at 9 months | Baseline, at nine months
  Number of words read (M)(standard deviation)
Change from baseline E index ( Alouatte-R test) at 9 months | Baseline, at nine months
  Number of errors (E)(standard deviation)
Change from baseline CM index ( Alouatte-R test) at 9 months | Baseline, at nine months
  Precision index (CM)(standard deviation)
Change from baseline CTL index ( Alouatte-R test) at 9 months | Baseline, at nine months
  Speed index (CTL)(standard deviation)
Change from baseline Regular ODEDYS test at 9 months | Baseline, at nine months
  Regular words reading, Screening tools for dyslexia (ODEDYS)(standard deviation)
Change from baseline Irregular ODEDYS test at 9 months | Baseline, at nine months
  Irregular words reading (standard deviation)
change from baseline Pseudo-words ODEDYS test at 9 months | Baseline, at nine months
  Pseudo-words reading (standard deviation)
Change from base line DFF VOG at 9 months | Baseline, at nine months
  Duration of first fixation (DFF), of the measured reading in Video Oculography (VOG),
Change from baseline DL VOG at 9 months | Baseline, at nine months
  Duration of look (DL), of the measured reading in Video Oculography (VOG),
Change from baseline TFT VOG at 9 months | Baseline, at nine months
  Total fixation time (TFT), of the measured reading in Video Oculography (VOG),
Observation of the evolution of the shape of maxwells spots from baseline at 9 months | Baseline, at nine months
  From the shape of Maxwell's tasks to the fovea-scope
Vertical orthophoria | Baseline, at nine months
  Comparison of the evolution of reading tests, taking into account the presence or absence of localization instability, whatever the treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Sparrow, MCF, Study Director — Scalab CNRS 9193, Lille University
Locations (1):
- Scalab CNRS 9193, Villeneuve-d'Ascq, Haut de France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quercia P, Quercia M, Feiss LJ, Allaert F. The distinctive vertical heterophoria of dyslexics. Clin Ophthalmol. 2015 Sep 25;9:1785-97. doi: 10.2147/OPTH.S88497. eCollection 2015. PMID 26445526